CLINICAL TRIAL: NCT07368595
Title: Comparison of Conjunctival Goblet Cell Density in Dry Eye Patients Treated With Cyclosporine 0.1% Dissolved in Perfluorobutylpentane (Vevye®) or Generic 0.05% Cyclosporine Emulsion for 8 Weeks
Acronym: CSAGCD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Harrow Inc (Industry)
Responsible Party: Principal Investigator, Steven Pflugfelder, Professor of Ophthalmology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-58336
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Laboratory perfoming goblet cell analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vevye® (Experimental): Cyclosporine dissolved in perfluorobutylpentane (Vevye®)
  Interventions: Drug: Vevye®
- Cyclosporine emulsion (Active Comparator): Cyclosporine emulsion
  Interventions: Drug: Cyclosporine emulsion

INTERVENTIONS:
Drug: Vevye® — cyclosporine 0.1% in perfluoroalkane vehicle
  Arms: Vevye®
Drug: Cyclosporine emulsion — cyclosporine 0.05% emulsion
  Arms: Cyclosporine emulsion

SUMMARY:
This goal of this clinical trial is to compare the effects of two approved cyclosporine eye drops that have different concentrations and vehicles on the number of mucus producing conjunctival goblet cells in patients with dry eye disease to learn which one causes the greatest increase.

The main questions it aims to answer are:

Does one drug cause a greater increase in goblet cells? How many weeks does it take to see the difference?

Participants will:

Use the eye drops every day for 2 months Visit the clinic once every 2 weeks for exams and tests

DETAILED DESCRIPTION:
Sixty participants with dry eye will be randomized to receive either cyclosporine 0.1% dissolved in perfluorobutylpentane (Vevye®) or 0.05% cyclosporine emulsion (generic Restasis®) to instill in their eyes twice a day for 60 days. The number of mucus producing goblet cells will be measured in the conjunctiva in both eyes by impression cytology. The percentage change in goblet cell number from baseline (before treatment ) at day 60 is the primary endpoint. Treatment groups will also be compared at days 14 and 30.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, 18 years of age or older at enrollment. 2. Have a history of DED, clinician diagnosed or patient reported, within the 6 months prior to the enrollment visit.

  3. Have both of these signs of DED in the same eye at the Enrollment (baseline) visit:
  1. Total cornea fluorescein staining score ≥ 3 based on the modified National Eye Institute (NEI) grading scheme.
  2. Total conjunctival lissamine green staining score ≥ 2 based on the modified NEI grading scheme. 4. Unanesthetized Schirmer test score ≥ 5 and < 15mm/5 min in at least 1 eye at the enrollment visit.

     5. A SANDE eye discomfort visual analog questionnaire score of ≥ 35 at the enrollment visit.

     6. Good general and ocular health, as determined by the investigator using medical history and ophthalmic examination.

     7. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

     8. Have given written informed consent prior to any study related procedures. 9. Able and willing to follow study instructions and likely to complete all required study visits as assessed by the investigator.

     Exclusion Criteria:
* Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Male or female, 18 years of age or older at enrollment.
2. Have a history of DED, clinician diagnosed or patient reported, within the 6 months prior to the enrollment visit.
3. Have both of these signs of DED in the same eye at the Enrollment (baseline) visit:

   1. Total cornea fluorescein staining score ≥ 3 based on the modified National Eye Institute (NEI) grading scheme.
   2. Total conjunctival lissamine green staining score ≥ 2 based on the modified NEI grading scheme.
4. Unanesthetized Schirmer test score ≥ 5 and < 15mm/5 min in at least 1 eye at the enrollment visit.
5. A SANDE eye discomfort visual analog questionnaire score of ≥ 35 at the enrollment visit.
6. Good general and ocular health, as determined by the investigator using medical history and ophthalmic examination.
7. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
8. Have given written informed consent prior to any study related procedures.
9. Able and willing to follow study instructions and likely to complete all required study visits as assessed by the investigator.

Exclusion Criteria:

Subjects meeting any of the following criteria at the enrollment visit will be excluded from entry into the study:

Ophthalmic:

1. History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, interfere with the interpretation of the study results or subject safety, such as: significant conjunctival scarring; pterygium or nodular pinguecula; conjunctivitis, or inflammation not associated with DED; clinically significant anterior blepharitis (Staphylococcal or Demodex).
2. Other significant ophthalmic disease requiring topical medication (e.g., glaucoma, ocular hypertension), or other ophthalmic disease which the investigator believes may interfere with study findings or interpretation.
3. History of ocular surgery within 1 year prior to the Screening visit, including punctal cautery, corneal refractive, or anterior segment surgeries (e.g., cataract surgery or any surgery creating limbal or corneal incisions).
4. History of corneal transplant in one or both eyes.
5. Diagnosis of recurrent, ongoing, or active ocular infection including, but not limited to herpes simplex or zoster, bacterial or fungal keratitis.
6. Use of contact lenses in either eye within 90 days prior to the enrollment visit or planned use during the study.
7. Punctal or intracanalicular plug present in either eyelid within 90 days prior to the enrollment visit or anticipated plug insertion or occlusion at any time during the study.
8. Regular use, as assessed by the investigator, of lid hygiene or heat masks within 14 days prior to the Enrollment visit or any planned use during the study.
9. Use of lid heating therapy (i.e., LipiFlow®, iLUX®, Thermal OneTouch, TearCare®) or Meibomian gland probing/therapeutic expression within 90 days prior to enrollment or anticipated during the study.
10. Use of Intense Pulsed Light (IPL) therapy on eyelids within 90 days prior to enrollment or anticipated during the study.
11. Use of artificial tears within 24 hours prior to enrollment or anticipated use during the study.
12. Use of any topical ocular cyclosporine A formulation (e.g., ocular cyclosporine [Restasis®, Cequa™, Vevye™, generics] within 1 year prior to enrollment. Use of lifitegrast [Xiidra®]), perfluorohexyloctane [Meibo™]), Tryptyr™, or any topical ocular corticosteroid, or any non-steroidal-anti-inflammatory agents within 90 days prior to enrollment or anticipated use during the study.
13. Use of topical ocular autologous serum/plasma within 90 days prior to the enrollment or anticipated use during the study.
14. Use of any topical ocular glaucoma medication within 30 days prior to enrollment or anticipated use during the study.
15. Regular use, as defined by the investigator, of any other topical ocular medication not listed in Exclusion 11, 12, 13 or 14 within 14 days prior to the enrollment visit or anticipated use during the study (e.g., eye whitening products [Visine®, Lumify®], topical ocular antibiotics, topical ocular antihistamines, mast cell stabilizers, presbyopia correcting drops [e.g., Vuity™].
16. Use of Tyrvaya™ (varenicline solution, nasal spray 0.03 mg) within 90 days prior to the enrollment visit or anticipated use during the study.
17. Use of oral medications for the treatment of severe DED and/or Meibomian gland disease such as oral pilocarpine, oral cevimeline, oral macrolides, oral tetracyclines or tetracycline derivatives, and oral retinoids within 30 days prior to enrollment or anticipated use during the study.
18. General/Systemic:

    Initiation, discontinuation, or change in dose of a systemic medication known to cause ocular drying (e.g., antihistamines or antidepressants) less than 30 days prior to enrollment or a change in dosage is anticipated during the study. Note: occasional short-term use of these medications, such as systemic antihistamines will be permitted, provided that use was not within 7 days prior to enrollment. Initiation, discontinuation, or change in dose of a systemic corticosteroid less than 60 days prior to the enrollment visit or a change in dosage is anticipated during the study. Note: Non-ocular topically applied corticosteroids (including topical creams, nasal sprays and inhalers) will be permitted during the study, and the dose is not required to be stable.
19. Initiation, discontinuation, or change in dose of a systemic immunomodulator (e.g., hydroxychloroquine, methotrexate, cyclosporine) less than 60 days prior to the enrollment visit or a change in dosage is anticipated during the study.
20. Use of an investigational product or device within 30 days prior to the Screening visit.
21. At the enrollment visit, at the investigator's discretion, have uncontrolled or severe:

    1. Systemic allergy
    2. Rhinitis or sinusitis
    3. Atopic dermatitis involving the eyelids
22. History or presence of significant systemic disease (i.e.: cardiovascular, pulmonary, hepatic, renal, hematologic, immunologic). Significant is defined as any disease that, in the assessment of the Investigator, would put the safety of the subject at risk through participation, or would prevent or confound protocol-specified assessments (e.g., severe rheumatoid arthritis, severe systemic lupus erythematosus, uncontrolled immunodeficiency disease, etc.).
23. Known allergies or sensitivity to the study interventions or study diagnostic agents, including sodium fluorescein, lissamine green, etc.
24. Pregnant at enrollment, currently breastfeeding or plans to become pregnant or breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 60 days
  Percentage change from baseline in goblet cell density at Day 60

SECONDARY OUTCOMES:
Secondary Outcome 1 | 60 days
  Change from baseline in goblet cell density at Day 60
Secondary Outcome 2 | 60 days
  Proportion of subjects with an increase in areas covered by goblet cells at Day 60
Secondary Outcome 3 | 60 days
  Proportion of subjects with increase in mean goblet cell density at Day 60
Secondary Outcome 4 | Days 14 and 30
  Change from baseline in goblet cell density at Days 14 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Pflugfelder, M.D., Principal Investigator — Baylor College of Medicine